#### The GlaxoSmithKline group of companies

| Division : Worldwide Development | |
|----------------------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for PET imaging study to investigate the biodistribution and clearance of a GSK3128349 in Healthy Volunteers.

Compound Number : GSK3128349

Effective Date : 06-MAR-2017

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol RES117169.
- This RAP is intended to describe the PET, safety and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the SAC deliverable.

#### **Author's Name and Functional Area:**

| PPD | | 06-MAR-2017 |
|-----------------|---------------------------------------|-------------|
| Senior Statisti | cian, Clinical Statistics (QSI) | 00-MAK-201/ |
| PPD | | 06-MAR-2017 |
| Systems Mode | elling and Translational Biology, PTS | 00-MAK-201/ |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# Reviewed by:

| PPD | 11-JAN-2017 |
|-----------------------------------|------------------|
| CPSSO, PCPS | 11-3/111-2017 |
| PPD | 06-MAR-2017 |
| Translational Medicine, PTS | 00 WITH 2017 |
| PPD | 06-MAR-2017 |
| Data Management | 00 WITH 2017 |
| PPD | 06-MAR-2017 |
| Clinical Programming, PCPS | 00-1417 114-2017 |
| PPD | 06-MAR-2017 |
| Project Manager, Clinical Imaging | 00-WAR-201/ |

The final RAP approval will be given by

# Approved Via E-mail by:

# Email approval on file

| PPD | Statistics & Programming, QSI | 06-MAR-2017 |
|-----|-------------------------------|-------------|
|-----|-------------------------------|-------------|

# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | REPORTING & ANALYSIS PLAN SYNPOSIS | 5 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 7<br>8 |
| 3. | PLANNED ANALYSES | 9 |
| 4. | ANALYSIS POPULATIONS | |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS | 11 |
| 6. | STUDY POPULATION ANALYSES | |
| 7. | PRIMARY STATISTICAL ANALYSES | 13<br>13<br>13 |
| 8. | SECONDARY STATISTICAL ANALYSES 8.1. Pharmacokinetic Analyses 8.1.1. Overview of Planned Pharmacokinetic Analyses 8.1.2. Drug Concentration Measures 8.1.3. Pharmacokinetic Parameters 8.1.3.1. Deriving Pharmacokinetic Parameters 8.2. Safety Analyses 8.2.1. Overview of Planned Adverse Event Analyses 8.2.2. Overview of Planned Clinical Laboratory Analyses 8.2.3. Overview of Planned Other Safety Analyses | 15<br>16<br>16<br>16<br>18<br>18 |
| 9. | REFERENCES | 21 |
| 10. | APPENDICES 10.1. Appendix 1: Protocol Deviation Management 10.1.1. Exclusions from Per Protocol Population 10.2. Appendix 2: Time & Events 10.2.1. Protocol Defined Time & Events 10.3. Appendix 3: Data Display Standards & Handling Conventions 10.3.1. Study Treatment & Sub-group Display Descriptors | 23<br>24<br>24 |


RES117169

| | 10.3.2. | Baseline D | efinition & Derivations | 26 |
|---|---|---|---|---|
| | | 10.3.2.1. | Baseline Definitions | 26 |
| | | 10.3.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | 26 |
| | 10.3.3. | Reporting | Process & Standards | 27 |
| 10.4. | Appendi | x 4: Derived | and Transformed Data | 29 |
| | 10.4.1. | General | | 29 |
| | 10.4.2. | Study Pop | ulation | 29 |
| | 10.4.3. | | | |
| 10.5. | Appendi | x 5: Premati | ure Withdrawals & Handling of Missing Data | 31 |
| | 10.5.1. | Premature | Withdrawals | 31 |
| | 10.5.2. | Handling o | f Missing Data | 31 |
| | | 10.5.2.1. | Handling of Missing Dates | 31 |
| | | 10.5.2.2. | Handling of Partial Dates | 32 |
| 10.6. | Appendi | | of Potential Clinical Importance | |
| | 10.6.1. | Laboratory | Values | 33 |
| | 10.6.2. | ECG | | 34 |
| | 10.6.3. | | | |
| 10.7. | | x 7 – Abbre | viations & Trade Marks | 35 |
| | 10.7.1. | Abbreviation | ons | 35 |
| | 10.7.2. | Trademark | S | 36 |
| 10.8. | Appendi | | Oata Displays | |
| | 10.8.1. | | ay Numbering | |
| | 10.8.2. | | nple Shell Referencing | |
| | 10.8.3. | | e [Priority] | |
| | 10.8.4. | • | ulation Tables | |
| | 10.8.5. | | S | |
| | 10.8.6. | | es | |
| | 10.8.7. | | kinetic Tables | |
| | 10.8.8. | | kinetic Figures | |
| | 10.8.9. | • | les | |
| | 10.8.10. | | JS | |
| | | | istings | |
| 10.9. | <b>Appendi</b> | x 9: Exampl | e Mock Shells for Data Displays | 49 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Pharmacology Study Report for study RES117169. |
| Protocol | This RAP is based on the original protocol (Dated: 23/MAY/2016) for study RES117169 (GlaxoSmithKline Document Number 2014N202021_00) |
| Primary<br>Objective | Evaluate biodistribution of 89Zr-GSK3128349 in regions of interest following IV administration to support future AlbudAb products and the development of a PBPK model. |
| Primary<br>Endpoint | <ul> <li>Quantitative parameters (including but not limited to <sup>89</sup>Zr-GSK3128349 concentration) derived from Positron Emission Tomography – Computer Tomography (PET-CT) data (e.g. Standardised Uptake Values (SUVs)<sup>a</sup>, volume of Regions Of Interest (ROI) to assess average and total uptake into regions of interest (e.g. liver, kidney, muscle, spleen, heart, lung, bladder, thymus – if feasible -,blood and bone).</li> </ul> |
| Secondary<br>Objectives | <ul> <li>Measure PK of 89Zr-GSK3128349 by whole blood, plasma and urine radiolabel detection to support future AlbudAb products and the development of a PBPK model.</li> <li>Measure PK of GSK3128349 by mass spectroscopy (MS) to support the development of a PBPK model.</li> <li>Measure dosimetry of 89Zr-GSK3128349 from PET scans and blood radioactivity</li> <li>Assess the safety and tolerability of 89Zr-GSK3128349.</li> <li>Investigate the presence and levels of anti-GSK3128349 antibodies, including pre- and post-dose.</li> </ul> |
| Secondary<br>Endpoint | <ul> <li>Whole blood, plasma and urine radioactivity concentrations and derived pharmacokinetic parameters, as data allows, based on blood, plasma and urine scintillation counting.</li> <li>Plasma concentrations and derived pharmacokinetic parameters.</li> <li>Compare plasma exposure assessments via different GSK3128349 mass Spectroscopy methods.</li> <li>Organ doses (mSv)</li> <li>Effective dose (mSv)</li> <li>Adverse events (AEs), serious adverse events (SAEs).</li> <li>Safety laboratory values, proteinuria, electrocardiograms (ECGs) and vital signs.</li> </ul> |
| Study<br>Design | <ul> <li>A single cohort of six to eight healthy male subjects.</li> <li>An open label, single centre, single drug study to investigate the biodistribution and pharmacokinetics of the AlbudAb platform scaffold protein GSK3128349.</li> <li>After completion of the first 2 subjects, dosimetry assessments will be performed and used to refine the radiation dose administered to subsequent subjects. This data may also be used to adjust the time post dose for PET scans performed on subsequent subjects.</li> <li>The total duration of a subject's participation is approximately 10 weeks, including the screening period of up to 28 days.</li> </ul> |
| Analysis<br>Populations | 'Screen Failures Population' comprises of all potentially eligible subjects who have signed the ICF and subsequently fail screening. |

| Overview | Key Elements of the RAP |
|---|---|
| | <ul> <li>'Safety Population' comprises of all subjects who receive a dose of 89Zr-GSK3128349.</li> <li>'PK Population' comprises of Subjects in the 'Safety' population for whom a PK sample was obtained and analysed, and/or for which a PET scan was completed.</li> <li>'All Screened Population' comprises of all subjects who were screened (or 'pre screened') for the trial, irrespective of whether they were enrolled or not. </li> </ul> |
| Hypothesis | There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives. |
| Primary<br>Analyses | <ul> <li>Descriptive statistics where appropriate, (i.e. n, arithmetic mean, geometric mean, standard deviation, minimum, median and maximum) will be calculated for all generated PET-CT imaging endpoints over time.</li> <li>Graphical displays will be produced over time for applicable PET-CT imaging endpoints.</li> <li>If analysed, all data will be listed, including unscheduled and/or repeat assessments.</li> <li>If data permits, further statistical analyses (i.e. mixed effects models) will be performed to estimate quantitative parameters in ROI over time from PET-CT following IV administration.</li> </ul> |
| Secondary<br>Analyses | <ul> <li>Whole blood and plasma concentrations time data of 89Zr-GSK3128349 and plasma concentrations time data of GSK3128349 will be analyzed by non-compartmental methods.</li> <li>As data permits, from the plasma concentration-time data, the following PK parameters may be determined as data permits: Cmax, Tmax, t1/2,AUC(0-t), AUC(0-∞), clearance, volume of distribution.</li> <li>Pharmacokinetic data will be presented in graphical and/or tabular form, summarized descriptively and listed.</li> <li>Dosimetry results as organ radiation doses and subject effective dose will be listed.</li> <li>Safety, tolerability and immunogenicity data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards.</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 23/MAY/2016).

# 2.2. Study Objective(s) and Endpoint(s)

| Ob | jectives | Endpoints |
|---|---|---|
| Pri | mary Objectives | Primary Endpoints |
| 1) | Evaluate biodistribution of 89Zr-GSK3128349 in regions of interest following IV administration to support future AlbudAb products and the development of a PBPK model. | Quantitative parameters (including but not limited to 89Zr-GSK3128349 concentration) derived from Positron Emission Tomography – Computer Tomography (PET-CT) data (e.g. Standardised Uptake Values (SUVs)a, volume of Regions Of Interest (ROI) to assess average and total uptake into regions of interest (e.g. liver, kidney, muscle, spleen, heart, lung, bladder, thymus – if feasible -, blood and bone). |
| Se | condary Objectives | Secondary Endpoints |
| 1) | Measure PK of 89Zr-GSK3128349<br>by whole blood, plasma and urine<br>radiolabel detection to support<br>future AlbudAb products and the<br>development of a PBPK model. | Whole blood, plasma and urine radioactivity concentrations and derived pharmacokinetic parameters, as data allows, based on blood, plasma and urine scintillation counting. |
| 2) | Measure PK of GSK3128349 by mass spectroscopy (MS) to support the development of a PBPK model. | <ul> <li>Plasma concentrations and derived pharmacokinetic parameters.</li> <li>Compare plasma exposure assessments via different GSK3128349 mass spectroscopy methods.</li> </ul> |
| 3) | Measure dosimetry of 89Zr-<br>GSK3128349 from PET scans and<br>blood radioactivity. | <ul><li>Organ doses (mSv)</li><li>Effective dose (mSv)</li></ul> |
| 4) | Assess the safety and tolerability of 89Zr-GSK3128349. | <ul> <li>Adverse events (AEs), serious adverse events (SAEs).</li> <li>Safety laboratory values, proteinuria, electrocardiograms (ECGs) and vital signs.</li> </ul> |
| 5) | Investigate the presence and levels of anti-GSK3128349 antibodies, including pre- and post-dose. | <ul> <li>Incidence of anti-GSK3128349 antibodies.</li> <li>Serum titres of anti-GSK3128349 antibodies.</li> </ul> |

## 2.3. Study Design



# 2.4. Statistical Hypotheses

There are no formal statistical hypotheses being tested, due to the exploratory nature of the study. Where applicable, an estimation approach will be adopted to evaluate the primary objectives.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

There are no formal interim analyses planned. However, the following in-stream data review is planned:

Following completion of the first two subjects' PET scans, the study team will evaluate the emerging PET-CT scan data for:

 Dosimetry to potentially refine the radiation dose estimates, and to identify other ROlfor further investigation, if required.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened | The All Screened population is defined as all subjects who were screened for the trial, irrespective of whether they were enrolled or not. | Screen Failure |
| Safety | Comprised of all subjects who receive a dose of 89Zr-GSK3128349. | <ul><li>Study Population</li><li>Safety</li></ul> |
| PK | Subjects in the 'Safety' population for whom a PK sample was obtained and analysed, and/or for which a PET scan was completed. | • PK |

#### NOTES:

 Please refer to Appendix 8: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.
  This listing will be based on data as recorded on the inclusion/exclusion page of the
  eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|--------------|--------------------------------------------------------------|
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| Section 10.2 | Appendix 2: Time & Events |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7 – Abbreviations & Trade Marks |
| Section 10.8 | Appendix 8: List of Data Displays |
| Section 10.9 | Appendix 9: Example Mock Shells for Data Displays |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 8: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Study Population | Data | Data Displays Generated | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition | Υ | | |
| Reasons for Screen Failure | | | Υ |
| Reasons for Subject Withdrawal | | | Υ |
| Planned and Actual Treatments | | | Υ |
| Protocol Deviations | | | |
| Important Protocol Deviations | | | Y |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Y [1] |
| Populations Analysed | · | | |
| Study Population | Υ | | |
| Subjects Excluded from Any Population | | | Υ |
| Demographic and Baseline Characteristics | · | | |
| Demographic Characteristics | Υ | | Υ |
| Race and Racial Combinations | Υ | | Y [2] |
| Race and Racial Combination Details | Y | | |
| Prior and Concomitant Medications | · | | |
| Medical Conditions (Current/Past) | Υ | | Υ |
| Concomitant Medication | Υ | | Υ |
| Exposure and Treatment Compliance | 1 | | 1 |
| Exposure to Study Treatment | | | Υ |
| NOTES - | 1 | 1 | L |

#### NOTES:

Y = Yes display generated.

<sup>[1]</sup> Listing also includes analysis population exclusions.

<sup>[2]</sup> Listing of race

#### 7. PRIMARY STATISTICAL ANALYSES

### 7.1. PET Analyses

# 7.1.1. Overview of Planned PET Analyses

The PET analyses will be based on the Pharmacokinetic population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 8: List of Data Displays.

Table 3 Overview of Planned PET Analyses

| [Endpoint / | | | | | | | |
|---|---|---|---|---|---|---|---|
| Parameter/ Display | Sta | ats An | alysis | Sum | mary | Individual | |
| Type] | T | F | L | T | F | F | L |
| Mean SUV | | | | Υ | Υ | Υ | Υ |
| Peak SUV | | | | Υ | Υ | Υ | Υ |
| Max SUV | | | | Υ | Υ | Υ | Υ |
| Activity Conc. Mean | | | | Υ | Υ | Υ | Υ |
| Total Activity | | | | Υ | | Υ | Υ |
| ROI Volume | | | | Υ | | | Υ |
| Percent Injected Dose | | | | Υ | Υ | Υ | Υ |
| Organ Doses | | | | Υ | Υ | | Υ |
| Effective Dose | | | | Υ | Υ | | Υ |

#### 7.1.2. PET Scan Parameters

#### 7.1.2.1. Deriving PET Scan Parameters

 The PET Scan parameters will be compiled into csv files as per specifications agreed in the External Data Vendor Agreement and will be transmitted to GSK via the External Alliance Portal

Table 4 Derived PET Scan Parameters

| Parameter | Parameter Description |
|---|---|
| SUV Mean | Ratio of tissue mean radioactivity concentration, averaged over a larger RoI, at a |
| - Tream | point in time C(T) and the injected dose of radioactivity per kilogram of the |
| | patient's body weight for larger regions of interest(>=3 cm): |
| | SUV = C(T)/[injection dose (MBq)/patient's weight (kg)] |
| SUV Peak | Ratio of tissue radioactivity concentration, averaged over a small sphere of defined |
| Tour | diameter (typically 10 mm) at a point in time C(T) and the injected dose of |
| | radioactivity per kilogram of the patient's body weight for smaller regions of |
| | interest: |
| | SUV = C(T)/[injection dose (MBq)/patient's weight (kg)] |
| SUV max | Ratio of maximum tissue radioactivity signal at a point in time C(T) and the |
| | injected dose of radioactivity per kilogram of the patient's body weight for larger |
| | regions of interest(>=3 cm): |
| | SUV = C(T)/[injection dose (MBq)/patient's weight (kg)] |

| Parameter | Parameter Description |
|---|---|
| Activity | Tissue mean radioactivity in Bq/ml from the RoI used for SUVmean |
| Conc. | |
| Mean | |
| Total | The total amount of radioactivity in MBq or Bq contained within ROI at time (T). |
| Activity | This corresponds to the total organ radioactivity if ROI corresponds to the total |
| | tissue volume. |
| ROI | The volume of the ROI used in measurements |
| Volume | |
| Percent | The percent of Injected dose found within ROI at time (T) |
| Injected | |
| Dose | |
| Organ | The amount of radiation delivered to a particular organ |
| Doses | |
| Effective | The tissue-weighted sum of the organ doses in all specified tissues and organs of |
| Dose | the human body |

## 7.1.2.2. Statistical Analysis of PET Scan Parameters

All derived PET Scan Imaging parameters will be summarized where appropriate, (i.e. n, arithmetic mean, standard deviation, minimum, median and maximum) over time. Graphical displays will also be produced over time for applicable PET-CT imaging endpoints.

Listings will be produced for all the collected data.

# 8. SECONDARY STATISTICAL ANALYSES

### 8.1. Pharmacokinetic Analyses

# 8.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the PK population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with full details being presented in Appendix 8: List of Data Displays.

 Table 5
 Overview of Planned Pharmacokinetic Analyses

| [Endpoint / | Untransformed | | | | | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| Type] | Τ | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| PK Concentration | | | | | | | | | | | | | | |
| Whole blood | | | | | <b>Y</b> [1] | <b>Y</b> [1] | Υ | | | | | | | |
| concentration of <sup>89</sup> Zr-<br>GSK3128349 | | | | Υ | | | | | | | | | | |
| Plasma Concentration of 89Zr-GSK3128349 | | | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Y | | | | | | | |
| Plasma concentration of GSK3128349 | | | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Y | | | | | | | |
| Urine Concentration of 89Zr-GSK3128349 | | | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Y | | | | | | | |
| PK Parameters | | | | • | • | | | | | | | | • | |
| Derived PK parameters | | | | Υ | | | Υ | | | | Υ | | | |
| for whole blood | | | | | | | | | | | | | | |
| concentration of 89Zr-<br>GSK3128349 | | | | | | | | | | | | | | |
| Derived PK parameters | | | | Υ | | | Υ | | | | Υ | | | |
| for plasma | | | | | | | | | | | | | | |
| concentration of <sup>89</sup> Zr-<br>GSK3128349 | | | | | | | | | | | | | | |
| Derived PK parameters | | | | Υ | | | Υ | | | | Υ | | | |
| for plasma | | | | | | | | | | | | | | |
| concentration of | | | | | | | | | | | | | | |
| GSK3128349 | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Y<sup>[1]</sup>= Linear and Semi-Log Plots would be produced

#### 8.1.1.1. **Analyses**

Whole blood and plasma concentrations time data of 89Zr-GSK3128349 and plasma concentrations time data of GSK3128349 will be analyzed by non-compartmental methods. From the plasma concentration-time data, the following PK parameters may be determined as data permits:

Maximum observed plasma concentration (Cmax), Time to achieve Cmax (Tmax), Apparent terminal phase half-life (t1/2), Area under the concentration-time curve from time zero (predose) to last time of quantifiable concentration within a subject (AUC[0-t]) for 89Zr-GSK3128349 and GSK3128349, Area under the concentration-time curve from time zero (predose) extrapolated to infinite time (AUC[0-∞]) only for GSK3128349, Clearance and Volume of distribution.

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively. Figures for individual plasma concentrations will be presented on both a linear and semilog scale for <sup>89</sup>Zr-GSK3128349 and GSK3128349. Linear and semi-log figures for mean and median plasma concentrations versus time for each treatment regimen will also be generated.

For each of the derived PK parameters of <sup>89</sup>Zr-GSK3128349 and GSK3128349, the following summary statistics will be calculated: n (number of observations), arithmetic mean, standard deviation, median, minimum, maximum, and the 95% confidence interval of arithmetic mean. In addition, summary statistics for log-transformed PK parameters [i.e., AUC(0-t), AUC(0-∞), Cmax, Clearance, t½ and Volume], except tmax will include geometric mean, 95% confidence interval of the geometric mean, standard deviation of the logarithmically transformed data, and inter-subject coefficient of variation [CVb (%)].

## 8.1.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).

#### 8.1.3. Pharmacokinetic Parameters

#### 8.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Matlab 2016b/SimBiology v5.4, Phoenix 6.3 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 5 will be determined from the 89Zr-GSK3128349 and GSK3128349 concentration-time data, as data permits.

 Table 6
 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t <sub>z</sub> ) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration $(C(\boldsymbol{t}_{z}))$ will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| | $AUMC(0-t_z) = \int_0^{t_z} C(t) \times dt$ |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: $AUC = AUC(Q - t) + \frac{C(t_z)}{lambda_z}$ |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: |
| | $t_{\frac{1}{2}} = \frac{\ln(2)}{lambda_{-}z}$ |
| lambda_z | The terminal phase rate constant |
| V_ss | Apparent volume of distribution at steady state $V_{SS} = \frac{Dose \times AUMC}{AUC^2}$ |
| AUMC | Total area under the first moment of the concentration—time curve extrapolating to Inf using lambda_z $AUMC = AUMC(O - t) + \frac{C(t_x)}{lambda_z^2} + \frac{t_x \times C(t_x)}{lambda_z}$ |
| AUMC(0-t <sub>z</sub> ) | Area under the first moment of the concentration—time curve from time 0 to the last time point $t_z$ . $AUMC(O - t_z) = \int_0^{t_z} t \times C(t) \times dt$ |
| MRT | Mean residence time. $MRT = \frac{AUMC}{AUC}$ |
| CL | Total drug clearance $CL = \frac{Dose}{AUC}$ |

# 1. NOTES:

Additional parameters may be included as required.

# 8.2. Safety Analyses

# 8.2.1. Overview of Planned Adverse Event Analyses

The safety analyses will be based on the Safety population, unless otherwise specified. This section will be completed in the final RAP.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 8: List of Data Displays.

Table 7 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | oint / Parameter/ Display Type Absolute | | |
|---|---|---|---|
| | Sun | Individual | |
| | T | L | |
| Adverse Events (AEs) | | | |
| All AEs by System Organ Class | Υ | | Y |
| All Drug-Related AEs by System Organ Class | Υ | | Y |
| Subject Numbers for Individual AEs | | | Y |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Serious AEs by System Organ Class | Υ | | Υ |
| Reasons for Considering as a Serious AE | | | Υ |
| AEs Leading to Withdrawal from Study | Υ | | Υ |

#### NOTES:

 T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.

# 8.2.2. Overview of Planned Clinical Laboratory Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 8: List of Data Displays.

Table 8 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumn | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Clinical Chemistry Parameters | Υ | | | Υ | | |
| Chemistry Data for Subjects with Abnormalities of Potential Clinical Concern | | | Y | | | |
| Chemistry Data Abnormalities of Potential Clinical Importance | | | Y | | | |
| Hematology | | | | | | |
| Hematology Parameters | Υ | | | Υ | | |
| Hematology Data for Subjects with Abnormalities of Potential Clinical Concern | | | Y | | | |
| Hematology Data Abnormalities of Potential Clinical Importance | | | Y | | | |
| Urinalysis | | | | | | |
| Urine Concentration Data | Υ | | Y | Υ | | |

# 8.2.3. Overview of Planned Other Safety Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 8: List of Data Displays.

Table 9 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Summary | | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | | | | |
| ECG Values by Visit | Υ | | | Υ | | |
| All ECG Values for Subjects with a Value of PCI | | | Υ | | | |
| ECG Values of PCI | | | Υ | | | |
| Abnormal ECG Findings | | | Y | | | |
| Vital Signs | | | | | | |
| Vital Signs by Visit | Υ | | | Υ | | |
| All Vital Signs for Subjects with Values of PCI | | | Y | | | |
| Vital Signs Values of PCI | | | Υ | | | |

# 9. REFERENCES

GlaxoSmithKline Document Number 2014N202021\_00 Study ID RES117169 An open label positron emission tomography (PET) imaging study using 89Zirconium labelled GSK3128349 to investigate the biodistribution and clearance of an albumin binding domain antibody (AlbudAb) GSK3128349 following single dose intravenous administration in healthy male subjects.MAY/2016

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 Appendix 1: Protocol Deviation Management | |
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 Appendix 3: Data Display Standards & Handling Conventions | |
| | <ul> <li>Study Treatment &amp; Sub-group Display Descriptors</li> </ul> |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Other RAP App | endices |
| Section 10.7 | Appendix 7: Abbreviations & Trade Marks |
| Section 10.8 | Appendix 8List of Data Displays |
| Section 10.9 | Appendix 9: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management

#### 10.1.1. Exclusions from Per Protocol Population

As detailed in Section 4.1, Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan and a listing of important Protocol Deviations will be provided.

A Per Protocol Population is not being defined for this study. However additional exploratory sensitivity summaries may be considered, if there are protocol deviations that may affect the primary PET endpoints. Any additional sensitivity summaries will be documented in the CSR.

# 10.2. Appendix 2: Time & Events

#### 10.2.1. Protocol Defined Time & Events

Screening up to 28 days prior **Procedures** to day 1 Informed Consent Χ Χ Demographics Eligibility Х Χ Full Physical Exam Medical/Medication/Drug/Alcohol Hx Χ 12-lead ECG (triplicate) Χ Χ Vital Signs Urine Drug/Alcohol Χ HIV, Hep B and Hep C Screen1 Х Haem/Chem/Urinalysis Tests/UPCR Χ Χ Concomitant Medication Review 1 If test performed within 3 months prior to first dose of study treatment, testing at screening is not required

Day 31 Day -20 ± Day of study Day 13 ± 1 day Day 1 Day 2 Day 4 Day 6 ±2 2 days days Pre-dose 1 hour 3 hours 6 hours 8 hours 24 hours Admission to Unit X Brief Physical Exam Χ Χg Medical/Medication/Drug/Alcohol Hx Χ 12-lead ECG Χf Х Χ Vital Signs Urine Drug/Alcohol Х Urinalysis Χ  $\mathbf{X}^{i}$ Χ Χ Spot Urine Protein/Creatinine ratio Χe X Haematology Χ Χ Χ Clinical chemistry Χ Randomisation Immunogenicity Blood Sample Х IV Infusion Dosing Χ PET imaging and co-localising CT Χ Χ (first subject)a PET imaging and co-localising CT Χ Χ Χ Χ (second subject)a PET imaging and co-localising CT (subsequent subjects)a, b Χ Χ PK Blood Sampling for MS Х Χ Χ Χ Χ Х Χ Χ Χ PK Blood Sampling for scintillation Χ Χ Χ Χ Χ Χ Χ Χ X countingh Bladder Voido Χ Urine Collection<sup>d</sup>

| Day of study | Day - | | Day 1 | | | Day 2 | Day 4 | Day 6 | Day 13 ± 1 day | Day<br>20 ±<br>2<br>days | Day 31<br>±2<br>days | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post dosing | | Pre-dose | 0 | 1 hour | 3 hours | 6 hours | 8 hours | 24 hours | | | | | |
| Adverse Event Review | | | | <b>←</b> | | | | | | | | · | |
| Concomitant Medication Review | | <del></del> | | | | | | | | | | | |
| Discharge | | | | | | | | Χ | | | | | |
| Outpatient Visit | | | | | | | | | Х | Χ | Х | Х | X |

- a. Each PET/CT scan must be preceded by heart rate and blood pressure assessments.
- b. For subsequent subjects (3rd and beyond) timings of PET scans will be based on data analysis from subjects 1 and 2 and may be carried out anytime between 1 and 10-12 days post injection. A maximum of 4 PET scans will be conducted in each subject.
- c. Pre-dose urine will not be retained.
- d. 24 hour urine collection. Total volume will be measured. Part of urine sample will be used for scintillation counting. An aliquot will be utilized for UPCR assessment and another stored for later MS PK analysis if required. Based on data from first 2 subjects, urine may be collected for longer than 24 hrs post dose for subsequent subjects.
- e. Aliquot from 24 hr collection sample, taken after 24 hr collection is complete.
- f. Triplicate measurement
- g. Prior to discharge
- h. Aliquot from MS PK blood sample
- Urine sample to be collected prior to discharge

Note: all time points are relative to start of infusion administration.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

#### 10.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporti | ng |
| Code | Description | Description | Order |
| А | 1 mg of Zirconium labeled<br>GSK3128349 | GSK3128349 | 1 |

#### 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

| Parameter | Study Assess | Study Assessments Considered As Baseline | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | | |
| Haematology | X | | | Screening |
| Chemistry | X | Х | | Day -1 |
| Urinalysis | X | Х | | Day -1 |
| ECG | X | | X | Day 1(Pre-Dose)[1] |
| Vitals | Х | | Х | Day 1(Pre-Dose)[1] |

#### NOTES:

[1] Mean of Day 1 (Pre-Dose) values will taken as baseline.

#### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 10.3.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | Software |
| The currently support the currently support to the currently suppo | pported versions of SAS software SAS 9.4 will be used. |
| Reporting Area | Reporting Area |
| HARP Server | : uk1salx00175 |
| HARP Area | : gsk3128349/res117169/final |
| QC Spreadsheet | QC Spreadsheet : gsk3128349/res117169/final/qc |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards | |
| Generation of RTF Files | |
| RTF files will be generated for all the tables | |

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

| Reporting Standards | |
|---|---|
| <b>Unscheduled Visits</b> | Unscheduled Visits |
| <ul> <li>Unscheduled visi</li> </ul> | its will not be included in summary tables. |
| <ul> <li>Unscheduled visi</li> </ul> | its will not be included in figures. |
| All unscheduled v | visits will be included in listings. |
| <b>Descriptive Summa</b> | ry Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Summary Statistics Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | acokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and [between and or within] geometric coefficient of variation (CVb/w (%)) will be reported.</li> <li>[1] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> </ul> |
| Parameters Not<br>Being Log<br>Transformed | Tmax |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. **General**

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### 10.4.2. Study Population

#### **Demographics**

#### Age

- Screening date will be used as a reference date for calculating age.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### 10.4.3. Safety

#### **ECG Parameters**

#### RR Interval

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

#### **ECG Parameters**

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the follow-up visit. The end of the study is defined as the last subject's last visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to</li> </ul> |
| | be missing data and should be displayed as such. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | Start or end dates which are completely missing (i.e. no year specified) will |
| | remain missing, with no imputation applied. |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | /I | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 10.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range | | Clinical Concern Range |
|---|---|---|---|---|
| | | Lower | Upper | |
| Absolute | | | | |
| | | > 450 | | |
| Absolute QTc Interval | | > 450 | ≤ 479 | |
| | msec | ≥ 480 | ≤ 499 | |
| | | ≥ 500 | | |
| Absolute PR Interval | msec | < 110 | > 220 | |
| Absolute QRS Interval | msec | < 75 | > 110 | |

# 10.6.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7 – Abbreviations & Trade Marks

# 10.7.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

# 10.7.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

HARP

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin
## 10.8. Appendix 8: List of Data Displays

## 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.8 | |
| PET | 2.1 to 2.8 | 2.1 to 2.7 |
| Pharmacokinetic | 3.1 to 3.7 | 3.1 to 3.9 |
| Safety | 4.1 to 4.13 | |
| Section | Listi | ings |
| ICH Listings | 1 to 23 | |
| Other Listings | 24 to | o 38 |

### 10.8.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

### NOTES:

### 10.8.3. Deliverable [Priority]

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.8.4. Study Population Tables

| Study Pop | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.1. | Safety | ES1 | Summary of Subject Disposition | | SAC |
| 1.2. | All<br>Screened | ES6 | Summary of Reasons for Screen Failure | | SAC |
| 1.3. | All<br>Screened | SP1 | Summary of Study Populations | | SAC |
| 1.4. | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.5. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.6. | Safety | DM6 | Summary of Race and Racial Combination Details | | SAC |
| 1.7. | Safety | MH1 | Summary of Current/Past Medical Conditions | | SAC |
| 1.8. | Safety | CM1 | Summary of Concomitant Medications | | SAC |

## 10.8.5. PET Tables

| PET: Ta | PET: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.1. | PK | PET1 | Summary of Mean SUV for Each Organ at All Time Points | | SAC |
| 2.2. | PK | PET1 | Summary of Peak SUV for Each Organ at All Time Points | | SAC |
| 2.3. | PK | PET1 | Summary of Max SUV for Each Organ at All Time Points | | SAC |
| 2.4. | PK | PET1 | Summary of Volume of Regions of Interest for Each Organ at All Time Points | | SAC |
| 2.5. | PK | PET1 | Summary of Percent Injected Dose for Each Organ at All Time Points | | SAC |
| 2.6. | PK | PET1 | Summary of Activity Concentration Mean for Each Organ at All Time Points | | SAC |
| 2.7. | PK | PET1 | Summary of Total Uptake values for Each Organ at All Time Points | | SAC |
| 2.8. | PK | PET1 | Summary of Organ And Effective Dose | | SAC |

# 10.8.6. PET Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.1. | PK | FIG1 | Individual Subject Single Panel Plot : Mean SUV over Time | Y-axis: Result X-axis: Planned Time Points | SAC |
| 2.2. | PK | FIG1 | Individual Subject Single Panel Plot : Peak SUV over Time | Y-axis: Result X-axis: Planned Time Points | SAC |
| 2.3. | PK | FIG1 | Individual Subject Single Panel Plot : Max SUV over Time | Y-axis: Result X-axis: Planned Time Points | SAC |
| 2.4. | PK | FIG2 | Mean Profile (mean +/- SE) Plot : Mean SUV over Time | Y-Axis: Mean +/- SE X-Axis: Time Points | SAC |
| 2.5. | PK | FIG2 | Mean Profile (mean +/- SE) Plot : Peak SUV over Time | Y-Axis: Mean +/- SE X-Axis: Time Points | SAC |
| 2.6. | PK | FIG2 | Mean Profile (mean +/- SE) Plot : Max SUV over Time | Y-Axis: Mean +/- SE X-Axis: Time Points | SAC |
| 2.7. | PK | FIG1 | Percent Injected Dose over time | Y-Axis : Percent Injected Dose X-axis : Time Points | SAC |

### 10.8.7. Pharmacokinetic Tables

| PK : Ta | PK: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 3.1. | PK | PK01 | Summary of Whole blood concentration of 89Zr-GSK3128349 Pharmacokinetic Concentration-Time Data | | SAC |
| 3.2. | PK | PK01 | Summary of Plasma Concentration of 89Zr-GSK3128349<br>Pharmacokinetic Concentration-Time Data | | SAC |
| 3.3. | PK | PK01 | Summary of Plasma Concentration of GSK3128349 Pharmacokinetic Concentration-Time Data | | SAC |
| 3.4. | PK | PK01 | Summary of Urine Concentration of 89Zr-GSK3128349<br>Pharmacokinetic Concentration-Time Data | | SAC |
| PK Para | ameters | | | | |
| 3.5. | PK | PK06 | Summary of Derived Pharmacokinetic parameters for whole blood concentration of 89Zr-GSK3128349(non-transformed and log-transformed) | | SAC |
| 3.6. | PK | PK06 | Summary of Derived Pharmacokinetic parameters for plasma concentration of 89Zr-GSK3128349(non-transformed and log-transformed) | | SAC |
| 3.7. | PK | PK06 | Summary of Derived Pharmacokinetic parameters for plasma concentration of GSK3128349(non-transformed and log-transformed) | | SAC |

## 10.8.8. Pharmacokinetic Figures

| PK : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration | | | | |
| 3.1. | PK | PK16a | Individual Whole Blood Concentration-Time Plots of 89Zr-GSK3128349 (Linear and Semi-log) | | SAC |
| 3.2. | PK | PK16a | Individual Plasma Concentration-Time Plots of 89Zr-GSK3128349 (Linear and Semi-log) | | SAC |
| 3.3. | PK | PK16a | Individual Plasma Concentration-Time Plots of GSK3128349 (Linear and Semi-log) | | SAC |
| 3.4. | PK | PK17 | Mean Whole Blood Concentration-Time Plots of 89Zr-GSK3128349 (Linear and Semi-log) | | SAC |
| 3.5. | PK | PK17 | Mean Plasma Concentration-Time Plots of 89Zr-GSK3128349 (Linear and Semi-log) | | SAC |
| 3.6. | PK | PK17 | Mean Plasma Concentration-Time Plots of GSK3128349 (Linear and Semi-log) | | SAC |
| 3.7. | PK | PK18 | Median Whole Blood Concentration-Time Plots of 89Zr-GSK3128349 (Linear and Semi-log) | | SAC |
| 3.8. | PK | PK18 | Median Plasma Concentration-Time Plots of 89Zr-GSK3128349 (Linear and Semi-log) | | SAC |
| 3.9. | PK | PK18 | Median Plasma Concentration-Time Plots of<br>GSK3128349 (Linear and Semi-log) | | SAC |

## 10.8.9. Safety Tables

| Safety : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 4.1. | Safety | CP_AE1p | Summary of All Adverse Events by System Organ Class | | SAC |
| 4.2. | Safety | CP_AE1p | Summary All Drug-Related Adverse Events by System Organ Class | | SAC |
| Labora | tory: Chemistry | 1 | | | |
| 4.3. | Safety | LB1 | Summary of Chemistry Data | | SAC |
| 4.4. | Safety | LB1 | Summary of Chemistry Changes from Baseline | | SAC |
| Labora | tory: Haematol | ogy | | | |
| 4.5. | Safety | LB1 | Summary of Haematology Data | | SAC |
| 4.6. | Safety | LB1 | Summary of Haematology Changes From Baseline | | SAC |
| Labora | tory: Urinalysis | | | | |
| 4.7 | Safety | LB1 | Summary of Urinalysis Data | | SAC |
| 4.8 | Safety | LB1 | Summary of Urinalysis Changes from Baseline | | SAC |
| ECG | | | | | |
| 4.9 | Safety | EG1 | Summary of ECG Findings | | SAC |
| 4.10 | Safety | EG2 | Summary of ECG values | | SAC |
| 4.11 | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | | SAC |
| Vital | Signs | | | | |
| 4.12 | Safety | VS1 | Summary of Vital Signs | | SAC |
| 4.13 | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit | | SAC |

# **10.8.10. ICH Listings**

| ICH : L | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | All Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| Protoc | ol Deviations | | | | |
| 3. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC |
| 4. | All Screened | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 5. | All Screened | SA3a | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 6. | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 7. | Safety | DM9 | Listing of Race | | SAC |
| Prior a | Prior and Concomitant Medications | | | | |
| 8. | Safety | CP_CM3 | Listing of Concomitant Medications | | SAC |
| Exposu | Exposure and Treatment Compliance | | | | |

| ICH : Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 9. | Safety | EX3 | Listing of Exposure Data | | SAC |
| Advers | e Events | | | | |
| 10. | Safety | CP_AE8 | Listing of All Adverse Events | | SAC |
| 11. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 12. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | <u> </u> |
| 13. | Safety | CP_AE8 | Listing of Serious Adverse Events | | SAC |
| 14. | Safety | | Listing of Reasons for considering as a Serious Adverse Event | | SAC |
| Chemis | stry Data | | | | <u>.</u> |
| 15. | Safety | LB5 | Listing of All Clinical Chemistry Data for Subjects with Abnormalities of Potential Clinical Importance | | SAC |
| 16. | Safety | LB5 | Listing of Chemistry Abnormalities of Potential Clinical Importance | | SAC |
| Labora | tory Data | | | | |
| 17. | Safety | LB5 | Listing of All Haematology Data for Subjects with Abnormalities of Potential Clinical Importance | | SAC |
| 18. | Safety | LB5 | Listing of Haematology Abnormalities of Potential Clinical Importance | | SAC |
| ECG | • | | | | , |
| 19. | Safety | CP_EG3 | Listing of All ECG Values for Subjects with a Value of Potential Clinical Importance | | SAC |
| 20. | Safety | CP_EG3 | Listing of ECG Values of Potential Clinical Importance | | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21. | Safety | CP_EG5 | Listing of Abnormal ECG Findings | | SAC |
| Vital S | Vital Signs | | | | |
| 22. | Safety | CP_VS4 | Listing of All Vital Signs for Subjects with Values of Potential Clinical Importance | | SAC |
| 23. | Safety | CP_VS4 | Listing of Vital Signs Values of Potential Clinical Importance | | SAC |

# 10.8.11. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 24. | PK | PK07 | Listing of Whole Blood Concentration Time Data of 89Zr-GSK3128349 | | SAC |
| 25. | PK | PK07 | Listing of Plasma Concentration Time Data of 89Zr-GSK3128349 | | SAC |
| 26. | PK | PK07 | Listing of Plasma Concentration Time Data of GSK3128349 | | SAC |
| 27. | PK | PK07 | Listing of Urine Concentration Time Data of 89Zr-GSK3128349 | | SAC |
| PK Para | ameters | | | | |
| 28. | PK | PK13 | Listing of Derived Pharmacokinetic Parameters for Whole Blood Concentration of 89Zr-GSK3128349 | | SAC |
| 29. | PK | PK13 | Listing of Derived Pharmacokinetic Parameters for Plasma Concentration of 89Zr-GSK3128349 | | SAC |
| 30. | PK | PK13 | Listing of Derived Pharmacokinetic Parameters for Plasma<br>Concentration of GSK3128349 | | SAC |
| PET | | | | | |
| 31. | PK | PET2 | Listing of Peak SUV Data | | SAC |
| 32. | PK | PET2 | Listing of Mean SUV Data | | SAC |
| 33. | PK | PET2 | Listing of Max SUV Data | | SAC |
| 34. | PK | PET2 | Listing of Activity Concentration Mean Data | | SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 35. | PK | PET2 | Listing of Volume of Regions of Interest | | SAC |
| 36. | PK | PET2 | Listing of Percent Injected Dose | | SAC |
| 37. | PK | PET3 | Listing of Organ Doses and Effective Doses | | SAC |
| Immunogenicity | | | | | |
| 38. | Safety | IMM2 | Listing of Immunogenicity Results | | SAC |

## 10.9. Appendix 9: Example Mock Shells for Data Displays

Example PET1

Protocol: RES117169 

Population: PK

Table X
Summary of Mean SUV for Each Organ At All Time Points[units]

| Organ | N | Planned<br>Relativ<br>e Time | n | Mean | 95% CI of Mean | SD | Media<br>n | Min | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Kidney | 24 | Pre- | 24 | XXXX.X | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | dose | | X | xxxx.xx) | X | X | X | |
| | | 30m | 24 | XXXX.X | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | | | X | xxxx.xx) | X | X | X | |
| | | 1h | 23 | xxxx.x | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | | | X | xxxx.xx) | X | X | X | |
| | | 2h | 24 | XXXX.X | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | | | X | xxxx.xx) | X | X | X | |
| Liver | 24 | Pre- | 24 | XXXX.X | (xxxx.xx, | XX.X | xxxx. | XXX | XXXX |
| | | dose | | X | xxxx.xx) | X | X | Х | |
| | | 30m | 21 | XXXX.X | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | | | X | xxxx.xx) | X | X | X | |
| | | 1h | 21 | XXXX.X | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | | | X | xxxx.xx) | X | X | X | |
| | | 2h | 21 | XXXX.X | (xxxx.xx, | XX.X | XXXX. | XXX | XXXX |
| | | | | X | xxxx.xx) | X | X | X | |


Example PET2

Protocol: RES117169

Population: PK

Listing X
Listing of Peak SUV Data

Planned

Inv./ Relative Date Actual Organ Result Subj. Visit Time Time (units)

PPD - This section has been excluded to protect patient privacy.


RES117169

Example PET3

Protocol: RES117169 

Population: PK

Listing X

Listing of Organ Doses and Effective Doses

Bone

Spleen Marrow Liver Lungs Kidney Body First Dose Subj. Treatment Age(y)/Sex (mSv) (mSv) (mSv) (mSv) (mSv) (mSv) GSK2849330

PPD - This section has been excluded to protect patient privacy.


RES117169

Example FIG1

Protocol: RES117169 

Population: PK

PPD - This section has been excluded to protect patient privacy.

Page 1 of 60

Individual Subject Single Panel Plot : PET Imaging Parameters over Time


Example FIG2

Protocol: RES117169

Population: PK

# Mean Profile (mean +/- SE) Plot : PET Imaging Parameters over Time

#### Treatment=A Test=Mean SUV Location=Kidney

